CLINICAL TRIAL: NCT02468414
Title: Safety & Efficacy of Prolonged Physiologic EPO Level Treatment of Anemia in ESRD Patients Undergoing Peritoneal Dialysis Using MDGN201 TARGTEPO
Brief Title: TARGTEPO Treatment for Anemia in PD US Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No statistical analysis was performed as only one subject was treated with MDGN201 TARGTEPO due to the Sponsor's decision to discontinue study.
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Collaborators: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-EP-RF-04
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Anemia of End Stage Renal Disease
Keywords: Peritoneal Dialysis; End Stage Renal Disease; Anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDGN201 TARGTEPO secreting EPO (Experimental): MDGN201 TARGTEPO secreting EPO
  Interventions: Biological: MDGN201 TARGTEPO

INTERVENTIONS:
Biological: MDGN201 TARGTEPO — MDGN201 TARGTEPO secreting EPO (18-25 IU/Kg/day)
Biological: MDGN201 TARGTEPO — MDGN201 TARGTEPO secreting EPO (35-45 IU/Kg/day)

SUMMARY:
The objectives of this study are to assess safety and to evaluate the biologic activity of TARGTEPO treatment in Peritoneal Dialysis patients

DETAILED DESCRIPTION:
This is a Phase II, open-label study. Each patient will be administered with a targeted dose of EPO delivered via TARGTEPO.

The targeted doses will be determined according to 2 cohorts as follows: Group A (18-25 IU/Kg/day), Group B (35-45 IU/Kg/day). The objective is to evaluate safety and biologic activity of TARGTEPO treatment when maintaining Hb levels within the target range of 9-12 g/dl. Biological activity assessments will include duration of TARGTEPO secretion as measured by serum EPO levels above baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects between 18 to 80 years of age at the time of screening visit.
2. Subject diagnosed with anemia due to Chronic Kidney Disease (CKD) Stage 5 on peritoneal dialysis treatment for at least 6 months. Average Hgb during last month between 9 to 12g/dL. Stable dose of ESAs over the past month prior to enrollment.
3. Hypertensive subjects are stable on anti HTN treatment for the past one month prior to enrollment and has Systolic blood pressure (BP) below 150 and Diastolic BP below 90 upon enrollment.
4. Kt/V > 1.
5. INR ≤ 1.2.
6. Serum albumin > 3.2.
7. Subjects with adequate iron stores (transferrin saturation > 20.0% and/or ferritin >100 ng/ml).
8. Capable of providing signed written informed consent to participate in the study.

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Subjects who receive oral anti-coagulation treatment (e.g. warfarin).
3. Subjects who receive acetylsalicylic acid (ASA) above 325 mg/day or patients who receive ASA treatment between 100mg/d and 325 mg/d who cannot discontinue it for 1 week prior to each Harvest or Implantation Procedure.
4. Congestive heart failure (New York Heart Association functional class III or IV).
5. Grand mal seizures within 2 years of the Screening Visit.
6. Clinical evidence of severe hyperparathyroidism as defined by parathyroid hormone (PTH) levels of > 10 times the upper normal limits.
7. Major surgery within 12 weeks of the Screening Visit.
8. Systemic hematologic diseases (e.g., sickle cell anemia, thalassemia (excluding thalassemia minor), myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia).
9. Current systemic infection, active inflammatory disease, or malignancy under active treatment.
10. Subjects known to have tested positive at any time in the past for antibodies to erythropoietic proteins.
11. Subject has history of malignancy within the past 2 years prior to the Screening Visit, with the exception of basal cell carcinoma.
12. Subjects with other concurrent severe and/or uncontrolled medical condition that could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive heart failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, uncompensated cirrhosis, active upper gastrointestinal (GI) tract ulceration).
13. Subject is currently enrolled in, or has not yet completed a period of at least 30 days or five half-lives of the investigational drug whichever is longer, since ending other investigational device or drug trial(s) prior to Screening Phase.
14. Psychiatric, addictive, or any other disorder that compromises ability to provide informed consent for participation in this study.
15. Female subjects of child-bearing potential and males that do not agree to use acceptable methods of contraception during the study.
16. Pregnant or lactating female subjects.
17. Chronic alcoholic or drug abuse subjects.
18. Steroid or other immunosuppressive treatment (other than topical or inhaled steroids).
19. Subjects unwilling or unable to comply with the study procedures.
20. EPO-naïve subjects.
21. Known sensitivity to gentamicin and amphotericin.
22. History of chronic or active hepatitis B and/or C infection or positive serology at screening, and known positive Human Immunodeficiency Virus (HIV) or positive serology at screening.
23. Subject had a blood transfusion within 84 days prior to Screening Visit.
24. Subject has a date for renal transplantation.
25. Refer to the United States Product Insert (USPI) - Depo-Medrol (DM) - Methylprednisolone Acetate - Injectable (Appendix A) for any concomitant drug taken by the patient, which its interactions with DM will warrant exclusion from this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, MD PhD, Study Chair — Medgenics Medical Israel Ltd.
Locations (1):
- Clinical Advancement Center, PLLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Early stage small feasibility study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 18-25 IU/Kg/day
- Group B: 35-45 IU/Kg/day
Period: Overall Study
Arm/Group | Group A | Group B
Started | 3 | 0
Successfully Screened | 2 | 0
Harvesting | 1 | 0
Implantation | 1 | 0
Safety Follow-up | 0 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Early Study Termination by Sponsor | 1 | 0
Not completed — Poor in-vitro secreting TARGTs | 1 | 0
Not completed — Screen Failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: TARGTEPO 18-25 IU/kg/day
- Group B: TARGTEPO 35-45 IU/kg/day
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Achieved Biological Activity of MDGN201 TARGTEPO Secretion as Measured by Serum EPO Levels Above Baseline.
Time Frame: 52 weeks
Population: No statistical analysis was performed as only one subject was treated with MDGN201 TARGTEPO due to the Sponsor's decision to discontinue study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=2) | Group B (N=0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=2) | Group B (N=0)
Local Contact Dermatitis, Right Upper Abdomen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute Viral Gasritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should the Primary Investigator (PI) wish to publish the results of this study, the PI agrees to provide the Sponsor with a manuscript for review 60 days prior to submission for publication. The Sponsor retains the right to delete from the manuscript information that is confidential and proprietary and to object to suggested publication and/or its timing (at the Sponsor's sole discretion).